CLINICAL TRIAL: NCT07187921
Title: Evaluation of a Finger Prick Collection Method for Measuring Alzheimer's Disease Blood Biomarkers (eDROP-AD)
Brief Title: Evaluation of a Finger Prick Collection Method for Measuring Alzheimer's Disease Blood Biomarkers
Acronym: eDROP-AD
Status: Completed | Type: Observational
Sponsor: Banner Health (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Other Study IDs: API-003; R01AG058468 (NIH)
Record Dates: First submitted 2025-09-11; First posted 2025-09-23 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Alzheimer Disease
Keywords: plasma pTau217
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — dried blood spot cards
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants who enrolled in Draw-10 and provided a venous blood sample

SUMMARY:
This is an observational study that will collect blood from a finger prick (Capitainer SEP10 single channel device) and assess the accuracy of pTau-217 testing in comparison to previously collected venous blood samples from the same individuals.

DETAILED DESCRIPTION:
Blood biomarkers offer a less invasive and cheaper method for identifying Alzheimer's disease (AD)-related pathophysiological changes. AD blood biomarkers are already being adopted by clinical practice and their use will only expand in coming years as access to AD modifying therapies increases. In addition, blood biomarkers are emerging as critical tools in AD research as they allow for streamlined identification of participants with the most relevant underlying levels of AD pathophysiology.

While blood tests offer a less invasive alternative to traditional detection methods (e.g., lumbar puncture, brain imaging), measuring biomarkers through venous blood draws can be logistically challenging, especially in resource-limited areas or for individuals unable to access specialized facilities. The use of blood collection cards could simplify the process, reduce the resources required, and make testing more accessible to a broader population. However, the accuracy of the measurement and their usability and tolerability to patients and research participants is not yet known. This study aims to evaluate acceptability of sampling using finger prick collection with a blood collection card for measuring pTau-217 as well as compare result accuracy to venous blood draw collection, thus addressing accessibility and scalability challenges in AD biomarker testing.

eDROP-AD is an ancillary study of the "Weekly blood draw study to understand the biological variability of plasma pTau-217" (Draw-10). Draw-10 is enrolling approximately 100 adults ages 50-80. Participants come to a study site weekly over a nine-week period for a venous blood draw with a phlebotomist. Participants at a select study site who provide a venous blood draw sample in Draw-10 will be invited to participate in eDROP-AD, leveraging the opportunity to evaluate the participant experience using blood collection cards and compare the results of the venous blood draw samples with blood samples acquired via the Capitainer SEP10 single channel device.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to provide informed consent for the eDROP-AD study.
* Enrolled in the Draw-10 study at Banner Alzheimer's Institute-Phoenix and provided at least one venous blood sample.
* Able and willing to fully comply with study procedures defined in this protocol.
* Written and spoken fluency in the English language.

Exclusion Criteria:

-

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Draw-10 study participants at Banner Alzheimer's Institute-Phoenix
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2025-09-29 (Actual); Primary Completion 2025-11-12 (Actual); Study Completion 2025-11-12 (Actual)

PRIMARY OUTCOMES:
Assess the accuracy of within-participant plasma pTau-217 testing on separated blood collected via finger prick with the Capitainer SEP10 single channel device in comparison to venipuncture-based collected samples. | Day 1
  compare pTau-217 assay value from finger prick blood sample to assay value from previously collected venipuncture-based collected blood
Characterize the feasibility of finger prick blood collection with the Capitainer SEP10 single channel device. | Day 1
  participant survey
Characterize the tolerability of finger prick blood collection with the Capitainer SEP10 single channel device. | Day 1
  participant survey
Characterize the acceptability of finger prick blood collection with the Capitainer SEP10 single channel device. | Day 1
  participant survey

SECONDARY OUTCOMES:
Analyze any differences in biomarker level from the finger prick blood samples collected via finger prick with the Capitainer SEP10 single channel device in comparison to venipuncture-based collected samples. | Day 1
  compare assay value from finger prick blood sample to assay value from previously collected venipuncture-based collected blood

CONTACTS AND LOCATIONS:
Overall Officials: Jessica B Langbaum, PhD, Principal Investigator — Banner Alzheimer's Institute
Locations (1):
- Banner Alzheimer's Institute, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
study dataset will be shared with qualified investigators
Supporting Information: Study Protocol, ICF
Time Frame: Data will be shared within 12 months after study completion